CLINICAL TRIAL: NCT02026245
Title: A Comparison of Two Electronic Goniometric Gloves in the Measurement of Joint Movement in Patients With Rheumatoid Arthritis
Brief Title: A Comparison of Two Electronic Gloves in the Measurement of Joint Movement in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulster (Other)
Collaborators: Western Health and Social Care Trust (Other)
Responsible Party: Principal Investigator, Dr Joan Condell, Senior Lecturer, University of Ulster
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: Dataglove-02
Record Dates: First submitted 2013-12-05; First posted 2014-01-01 (Estimated); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Rheumatoid Arthritis
Keywords: Arthritis; rheumatoid; joints; swelling; measurement; movement; electronic; data; glove; goniometry; outcome; stiffness
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 5DT electronic data glove (Experimental): Using the electronic data gloves to perform a set routine of movements.
  Intervention: Data gloves to perform movements
  Interventions: Device: Data gloves to perform movements
- Tyndall/UU electronic data glove (Experimental): Using the electronic data gloves to perform a set routine of movements
  Intervention: Data gloves to perform movements
  Interventions: Device: Data gloves to perform movements

INTERVENTIONS:
Device: Data gloves to perform movements — Using the electronic data gloves to perform a set routine of movements:
  * 5DT 'dataglove 14 Ultra' Electronic glove (commercially available)
  * New 'Tyndall/UU' developmental dataglove
  Other Names: 5DT; Tyndall/UU dataglove

SUMMARY:
In this study we will compare two electronic goniometric gloves to see if they can be used in research on joint movement in arthritis.

One of the gloves we will use is the commercially available '5DT Ultra 14 glove', the other is a glove that we have specially designed and developed for use in people with arthritis. Both gloves are 'high-end' gloves with sensors for all of the finger and thumb joints.

We aim to find out if the gloves are accurate and if they can be worn and used without too much discomfort by people with arthritis.

DETAILED DESCRIPTION:
This is an open pilot study to assess the usability and accuracy of two electronic goniometric gloves in measuring finger joint movement in patients with Rheumatoid Arthritis.

We will use questionnaires to assess pain, stiffness and disability. We will be using an inner disposable glove worn under the electronic goniometric gloves as this will be important for infection control in clinical use.

We will calibrate the electronic goniometric gloves using wooden blocks at predefined angles using our own software calibration process to optimise the accuracy of the glove for the individual patient.

The patient will flex and extend their fingers repeatedly to get measurements of the minimum and maximum angle of flexion in their joints. During these movements we will also capture the dynamic characteristics of movement such as maximum velocity. In this study a laptop will be used to capture and record all of the measurements from the electronic goniometric glove and record the time at which the measurements were taken.

Each electronic goniometric glove will be refitted for a second set of tests to assess variability due to the fitting process. We will record a full set of data from each set of movements for later analysis.

Finally, we will assess usability and establish if patients have a preference between the two electronic goniometric gloves.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 18 to 80
* Diagnosis of Rheumatoid arthritis
* Patients who have significant pain and stiffness in their hands
* Correct hand size to achieve a good fit to the electronic goniometric glove

Exclusion Criteria:

* Poor fit for the disposable surgical glove
* Severe pain in the right hand
* Severe swelling in the right hand (rated as such by the investigator)
* Major permanent deformities in the right hand
* Active hyperextension >30 degrees in any joint of the right hand
* Broken or infected skin in the right hand
* Known to have tested positive for Methicillin resistant staphylococcus aureus (MRSA) skin infections in the past
* Unable to don the lining disposable glove without significant discomfort
* History of Latex allergy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
The accuracy of joint angle measurement by each electronic goniometric glove will be compared with the accuracy of manual goniometry. | 1 day
  The standard error of measurement for each electronic goniometric glove will be used to evaluate the reliability of each electronic goniometric glove. This will be compared to the standard error of measurement for manual goniometry.

SECONDARY OUTCOMES:
The variability in the measurement of joint movement velocity | 1 day
  With rapid repeated movements of finger flexion and extension, the measured maximum velocity of movement should remain fairly constant. The intraclass correlation coefficient will be used to assess the variability in the measurement of joint movement velocity.
Variability of joint angle measurements by the electronic goniometric gloves will be assessed | 1 day
  The Intraclass Correlation coefficient for joint angle measurement will be measured for each electronic goniometric glove
The number of patients who withdraw or refuse to continue | 1 day
  Electronic goniometric gloves may not be easy to don and doff in patients with arthritis, particularly if used with an inner disposable glove. Because of the small numbers we will not apply a statistical analysis
Variation in joint angle movement between fit and refit | 1 day
  If a electronic goniometric glove relies on accurate sensor positioning, refitting may give widely varying results. Each glove will be refitted once.
Variation in joint angle measurement across the range of movement | 1 day
  With use of electronic goniometric gloves, joint angle measurement may be less accurate at the extremes of movement
Variation in joint angle movement across sensors - between digits | 1 day
  Although it may be assumed that the sensors in each digit should perform equally well, the movement of the stretch sensors over the joints may vary between digits. This analysis will test for this variability
The number of patients who prefer one electronic goniometric glove over the other | 1 day
  We will ask the patient which electronic goniometric glove they prefer. This will assess usability factors such as comfort, neatness of fit, and ease of donning and doffing.
The variation in joint angle measurement with force applied | 1 day
  We will use the Intra class correlation test to determine if the accuracy of measurements is affected by the patient gripping tightly against a moulded object held in the palm of their hand.
We will test the variability of joint angle measurements in wrist extension/flexion | 1 day
  We will compare the Intraclass Correlation coefficient for joint angle measurements carried out using the electronic goniometric glove in wrist extension/flexion

CONTACTS AND LOCATIONS:
Overall Officials: Philip Gardiner, MB BCh MD, Principal Investigator — WHSCT
Locations (1):
- Western Health and Social Care Trust, Londonderry, United Kingdom

IPD SHARING:
Plan to Share IPD: No
IPD may be considered available at a later date, anonymised.